CLINICAL TRIAL: NCT06594289
Title: Evaluation of the Safety and Effectiveness of Pringle Method Combined With IVC Flow Limiting and Blocking Method in Laparoscopic Hepatectomy Based on Non-restrictive Fluid Therapy Strategy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYSKY-2024-462-02
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Liver Tumor
Keywords: Liver cancer; Laparoscopic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Complete random grouping method was used in this study. Patients meeting the inclusion criteria were assigned to group A and Group B in a 1:1 ratio with 110 cases in each group by random number table method. The results are hidden in an opaque sealed envelope, which is then stored by the clinical study designer (i.e., a random code sheet). The researcher opened the envelope on the morning of the operation to obtain the group of patients and informed the operating physician and anesthesiologist to intervene accordingly according to the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group A (Pringle method + restricted fluid management + use of vasoactive drugs by anesthesiologists) : The means of use and anesthetic drugs in this group were all conventional technical means without special intervention, so it was the control group.
- Observation group (Experimental): Group B (Pringle method +IVC flow limiting and blocking method + open fluid intake during operation; Observation group: Patients in this group did not use anesthesia related drugs to control CVP, so they should strictly communicate with the anesthesiologist, and achieve homogeneity in the use of vasoactive drugs and narcotic drugs.
  Interventions: Procedure: In laparoscopic hepatectomy, the subhepatic inferior vena cava was restricted and the patient was given non-restricted intraoperative fluid intake

INTERVENTIONS:
Procedure: In laparoscopic hepatectomy, the subhepatic inferior vena cava was restricted and the patient was given non-restricted intraoperative fluid intake — The specific steps of IVC blocking were performed by the principal physician under laparoscopic operation: slightly incision of the posterior peritoneum on both sides of the inferior vena cava above the level of the renal vein. The "blood vessel blocking band" is passed behind the inferior vena cava on the left or right side of the inferior vena cava. According to the intraoperative situation, the blocking band (flow limiting blocking/incomplete blocking of subhepatic inferior vena cava) was tightened to control the bleeding from hepatic vein on the liver section. Patients in this group did not use vasoactive drugs/underuse means to control CVP, so they need to strictly communicate with the anesthesiologist, and take the fluid intake based on the physiological requirements and fluid loss of individual patients (cancel the restriction of fluid intake).
  Arms: Observation group

SUMMARY:
The relevant data of 220 patients undergoing laparoscopic hepatectomy in our hospital were collected. Based on randomization, blindness and inclusion and exclusion criteria, the patients were divided into group A (which included Pringle method + restricted fluid management + vasoactive drug use by anesthesiologists) and group B (which included: Pringle method +IVC flow limiting and blocking method, intraoperative fluid rehydration according to physiological requirements and expected loss, no or less vasoactive drugs used during the operation), and intraoperative and postoperative relevant indicators were compared between the two groups, such as; CVP value, fluctuation range, length of operation, time of liver amputation, total blood loss, amount of liver amputation, amount of blood transfusion, and amount of fluid perfusion. Internal environmental indicators: albumin, alanine aminotransferase, aspartate aminotransferase, γ-gt, total bilirubin, renal function, lactic acid, blood gas analysis (three times during the operation). Postoperative indexes: average length of stay and unplanned reoperation rate. While taking into account the safety, effectiveness and interpretability of statistical results, a new laparoscopic hepatectomy technique based on the optimized CLCVP process was constructed to control intraoperative bleeding and GDFT standardized and streamlined intervention strategy. This is not only an important innovation of the CLVCP concept, but also an important link to accelerate the implementation of laparoscopic liver resection technology in grassroots hospitals, and will significantly improve the quality of medical services, which can bring more accurate and efficient treatment programs to patients.

DETAILED DESCRIPTION:
Overall design Research hypothesis: Based on the non-restrictive fluid management strategy (intraoperative fluid rehydration according to physiological requirements and expected loss, no or less use of vasoactive drugs during the operation) combined with Pringle method and IVC flow restriction blocking method, the method of blocking hepatic blood flow was applied to effectively control intraoperative bleeding. Reduce the degree of intraoperative anesthesiologist dependence, improve the intraoperative compatibility between surgeons and anesthesiologists, and optimize the traditional CLVCP process, so as to achieve the goal of accurate maintenance of patients' organs in functional surgery and more rapid and widespread promotion of laparoscopic liver resection technology.

Type of study: A prospective randomized controlled study will be used in this study 5.2 Research and design process 5.2.1 Study the specific implementation process A total of 220 patients undergoing elective laparoscopic partial hepatectomy were selected from our hospital. All patients and their families knowingly and voluntarily signed informed consent before enrollment. On the basis of randomization and inclusion and exclusion criteria, the patients were divided into group A (110 cases) (Pringle method + restricted fluid management + use of vasoactive drugs by anesthesiologists) and group B (110 cases) (Pringle method +IVC flow restriction blocking + open fluid intake during the operation, and no/less use of vasoactive drugs during the operation). Intraoperative and postoperative related indexes were compared between the two groups, such as; CVP value, duration, fluctuation range, length of operation, time of liver amputation, total blood loss, amount of liver amputation, amount of blood transfusion, amount of liquid perfusion, three blood gas analysis during the operation, blood glucose, and dosage of vasoactive drugs. 3 days after operation: albumin, alanine aminotransferase, aspartate aminotransferase, gamma-GT, total bilirubin, renal function, lactic acid and other related indexes. Postoperative hospital stay (d), tracheal intubation and extubation time (d), surgical cost (ten thousand yuan), abdominal effusion, pulmonary infection, postoperative flatulence time (d), postoperative exhaust time (d), incision infection, intestinal obstruction. To comprehensively evaluate the safety and efficacy of Pringle method and IVC flow limiting blockade in the implementation of non-restrictive fluid intake strategies.

Ways to reduce bias

1. Complete random grouping: This study adopts the complete random grouping method; Patients meeting the inclusion criteria were assigned to group A and Group B in a 1:1 ratio with 110 cases in each group by random number table method. The results are hidden in an opaque sealed envelope, which is then stored by the clinical study designer (i.e., a random code sheet). The researcher opened the envelope on the morning of the operation to obtain the group of patients and informed the operating physician and anesthesiologist to intervene accordingly according to the study protocol.
2. Baseline control of patients Group A (Pringle method + restricted fluid management + use of vasoactive drugs by anesthesiologists) : The means of use and anesthetic drugs in this group were all conventional technical means without special intervention, so it was the control group.

Group B (Pringle method +IVC flow limiting and blocking method + open fluid intake during operation; Observation group: Patients in this group did not use anesthesia related drugs to control CVP, so they should strictly communicate with the anesthesiologist, and achieve homogeneity in the use of vasoactive drugs and narcotic drugs.

In order to reduce the deviation: 1. During the implementation of the subject, the group concealization was strictly implemented, and the designer informed the operating physician and anesthesiologist of the patient intervention plan one day before the operation.

2. Fluid intake 12 hours before surgery for all enrolled patients was strictly regulated according to preoperative ERAS.

3. All enrolled patients were strictly defined for the use of vasoactive drugs during the operation to reduce the deviation of statistical results caused by the use of different vascular drugs 4. All enrolled patients were performed by the same surgeon and anesthesiologist 5.4 Definition of the end of the study (e.g., the last study subject completes the last follow-up) The end of the study was defined when all enrolled patients completed surgery and the last patient completed follow-up 5.5 Statistical Analysis 5.5.1 Sample size and calculation basis Clinical data of patients undergoing laparoscopic hepatectomy in the Department of Hepatobiliary Surgery of Sun Yat-sen Memorial Hospital meeting the above inclusion criteria were collected. Intraoperative blood loss and intraoperative CVP control were used as the main observation indexes.

In this study, intraoperative blood loss and intraoperative CVP were respectively used to calculate the minimum sample size. According to previous observations, the mean difference of intraoperative blood loss between the two groups was about 28ml, the common standard deviation was conservatively estimated to be 55ml, the mean difference of intraoperative CVP between the two groups was about 2cmH2O, and the common standard deviation was conservatively estimated to be 1.5cmH2O. The Class I error α and class II error β of hypothesis test were set as 0.05, and the number of subjects in the two groups was 1:1. The PASS15.0 software was used for calculation, and the sample size of intraoperative blood loss was obtained as n=83 persons in each group, and the sample size of intraoperative CVP was obtained as n=13 persons in each group, and the larger value was adopted, that is, the sample size was 83 persons in each group. Assuming a 20% loss rate, the final sample size is 104 people per group, for a total of 208 people.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative Child-Pugh classification of liver function Grade A and grade B;
2. No contraindications for laparoscopic hepatectomy;
3. Liver diseases include: primary liver cancer, hepatic hemangioma, intrahepatic bile duct calculus, intrahepatic bile duct cell carcinoma, etc.
4. Patients voluntarily participate and sign informed consent;
5. According to the Ban difficulty scoring system of laparoscopic hepatectomy, patients with difficulty score of 5 or more were included; Neoplasms near the hepatic portal; Extensive hepatectomy (3 hepatic segments). Patients aged 18-70 years (including 18-70 years)

Exclusion Criteria:

1. Poor liver reserve function, ICG retention rate > 15%;
2. severe heart and lung diseases, unable to tolerate general anesthesia surgery;
3. Previous history of liver surgery;
4. More than medium amount of chest and abdominal fluid with clinical symptoms:
5. hepatic encephalopathy;
6. having a history of psychotropic drug abuse, unable to quit or having a history of mental disorders;
7. Patients who have received solid organ transplantation or bone marrow transplantation, or within 2 years before surgery
8. An active autoimmune disease requiring systemic treatment has occurred;
9. There is an immune deficiency disease or HIV infection;
10. Those who were not considered suitable for inclusion by the researchers.
11. Progression of the disease or toxic side effects or serious adverse events that the subjects could not tolerate before surgery after treatment;
12. Poor patient compliance, non-cooperation, concealment, false reporting and other phenomena: others
13. Cases where the principal investigator determines that the research protocol is seriously violated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Up to approximately 20 months：September 2024 - May 2026
  The amount of intraoperative blood loss is an important index to evaluate surgical safety
Intraoperative central venous pressure | Up to approximately 20 months：September 2024 - May 2026
  Central venous pressure is an important factor in the evaluation of blood loss after subhepatic inferior vena cava occlusion

SECONDARY OUTCOMES:
Level of aminotransferase | Up to approximately 20 months：September 2024 - May 2026
  An important indicator of liver function
level of Lactic acid | Up to approximately 20 months：September 2024 - May 2026
  An important indicator of liver and kidney metabolic function
Blood Sugar level | Up to approximately 20 months：September 2024 - May 2026
  An important indicator of liver synthesis
level of creatinine | Up to approximately 20 months：September 2024 - May 2026
  An important indicator of kidney function

OTHER OUTCOMES:
Postoperative complications, such as bile leakage, laparoscopic infection, deep vein thrombosis of the lower extremity, and unplanned re-entry surgery | Up to approximately 20 months：September 2024 - May 2026
  Indicators to evaluate postoperative safety

CONTACTS AND LOCATIONS:
Overall Officials: Yajin Chen, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China/Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
After the paper is published, you can contact us through the corresponding author's email address. We are willing to share the data results